CLINICAL TRIAL: NCT05421299
Title: Overall Survival in 7/8 HLA-Matched Hematopoietic Stem Cell Transplantation Patients Treated With Abatacept Combined With a Calcineurin Inhibitor and Methotrexate- An Analysis of the Center for International Blood and Marrow Transplant Research (CIBMTR) Database
Brief Title: A Study to Assess 7/8 HLA-matched Hematopoietic Stem Cell Transplantation Participants Treated With or Without Abatacept in Combination With a Calcineurin Inhibitor and Methotrexate
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-841
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Stem Cell Transplantation
Keywords: Abatacept; Orencia; Hematopoietic Stem Cell Transplantation (HSCT); aGVHD Prophylaxis; Unrelated Donor; Mismatched Donor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Abatacept Group: Participants with acute myeloid leukemia (AML), acute lymphoblastic leukemia (ALL), chronic myelogenous leukemia (CML), myelodysplastic syndromes (MDS), hodgkin lymphoma (HL), or non-hodgkin lymphoma (NHL) who have a bone marrow (BM) or peripheral blood (PB) stem cell donor who is HLA-matched at 7/8 loci (A, B, C, DRB1) who received abatacept.
- Comparator Group: Participants with AML, ALL, CML, MDS, HL, or NHL who have a BM or PB stem cell donor who is HLA-matched at 7/8 loci (A, B, C, DRB1) who did not receive abatacept.

SUMMARY:
The purpose of this study is to estimate overall survival (OS) for participants treated with abatacept versus those not treated with abatacept prior to hematopoietic stem cell transplantation (HSCT). Participants were included if their donors were unrelated and had 1-allele mismatched human leukocyte antigen (HLA) status.

ELIGIBILITY:
Inclusion Criteria:

* Participants who underwent first allogenic transplant in the US
* Participants with an unrelated donor who are HLA-matched at 7/8 loci (A, B, C, DRB1)
* Participants at least 6 years old with weight at least 20 kilograms
* Participants with a Karnofsky/Lansky Performance Score ≥80%
* Participants whose first allogeneic transplant occurred from January 1, 2011 to December 31, 2018
* Participants with any of the following diseases: AML, ALL, CML, MDS, HL, NHL
* Participants with any of the following graft versus host disease (GVHD) prophylaxis treatments:
* CNI plus MTX (with or without ATG and with or without abatacept); or
* Post-transplant cyclophosphamide (PT-Cy) without antithymocyte globulin (ATG)
* Participants treated with any of the following conditioning regiments: total body irradiation (TBI)/cyclophosphamide (Cy), busulfan (Bu)/Cy, Bu/fludarabine (flu), Flu/Melphalan (MEL)

Exclusion Criteria:

* Participants with missing information on ATG (yes/no)
* Participants receiving alemtuzumab (Campath)
* Participants with cord blood grafts
* Participants with non-MDS myeloproliferative disorders (NOTE: Participants with chronic myelomonocytic leukemia [CMMoL] will be included)
* Participants who did not consent to participate in research
* Participants treated at embargoed centers for research
* Participants treated with abatacept and ATG
* Among non-abatacept treated participants, participants transplanted at centers with abatacept trial participants
* Participants with any of the following missing propensity score variables:
* Disease status at transplantation (early, intermediate, advanced HL and NHL-chemosensitive)
* Age
* Gender (male, female)
* HSCT graft source (bone marrow [BM], peripheral blood [PB])
* Conditioning intensity (myeloablative, non-myeloablative / reduced intensity)
* Karnofsky/Lansky Performance Score (80%, 90-100%)
* CNI type (tacrolimus, CsA)

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study uses data routinely collected into the Center for International Blood and Marrow Transplant Research (CIBMTR) database. From the patterns of use analysis of the CIBMTR database, the majority of participants who received calcineurin inhibitor (CNI) plus methotrexate (MTX) plus abatacept were treated between 2011 and 2018. The study population has been selected to approximate the inclusion and exclusion criteria of the ABA2 clinical trial as closely as possible.
Sampling Method: Non-Probability Sample
Enrollment: 378 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Overall Survival in 7/8 HLA-matched Participants Treated with Study Therapy | Up to 180 days post transplant

SECONDARY OUTCOMES:
Overall Survival in Participants Treated with Study Therapy | Up to 180 days post transplant
Overall Survival in Participants Treated with Study Therapy Plus Tacrolimus | Up to 180 days post transplant

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Princeton, New Jersey, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html